CLINICAL TRIAL: NCT00468013
Title: A Computer-Based Intervention for Medically Unexplained Physical Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P15-MUPS-8484
Record Dates: First submitted 2007-04-27; First posted 2007-05-01 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Fibromyalgia; Irritable Bowel Syndrome; Chronic Fatigue Syndrome
Keywords: Fibromyalgia; Irritable Bowel; Chronic Fatigue; Medically Unexplained Symptoms; Resilience Building Exercises; Depression; Well-Being
MeSH Terms: conditions — Fibromyalgia; Irritable Bowel Syndrome; Fatigue Syndrome, Chronic; Medically Unexplained Symptoms; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Computer-based exercises to be executed at home.
  Interventions: Behavioral: Resilience Building Exercises
- 2 (Sham Comparator): Computer-based exercises to be executed at home.
  Interventions: Behavioral: Journaling

INTERVENTIONS:
Behavioral: Resilience Building Exercises — Weekly exercises for 6 weeks
  Arms: 1
Behavioral: Journaling — Weekly exercises for 6 weeks
  Arms: 2

SUMMARY:
In this study 60 people with medically unexplained physical symptoms (MUPS) will receive either a 6-session resilience skill building intervention provided fully online or a weekly computerized journaling assignment. Both programs can be completed from home. Participants will complete questionnaires both before and after the intervention and changes in symptoms, mood and satisfaction with life will be assessed.

DETAILED DESCRIPTION:
SUBJECTS: Sixty patients between the ages of 18 and 80 will be recruited from primary care clinics affiliated with the University of Medicine and Dentistry of New Jersey - Robert Wood Johnson Medical School (UMDNJ-RWJMS). Qualified patients will be primary care patients who meet the following inclusion and exclusion criteria: Patients between the ages of 18 and 75 seeking medical care for physical symptoms (i.e., persistent fatigue, pain complaints, and gastrointestinal, cardiovascular or musculoskeletal symptoms). No major medical illness to explain symptom(s) is found after detailed physical and laboratory assessment. Patients with common disorders such as hypertension, asthma, diabetes, low back strain, etc., will be included if in the opinion of the physician the presenting physical symptoms are not due to the underlying disorder. In order to enter the study, patients must meet criteria for at least 4 medically unexplained symptoms out of the 42 somatic symptoms listed in the Composite International Diagnostic Interview (CIDI) rated as currently present if males and at least 6 symptoms if females (Escobar's abridged criteria). Patients without ready access to a computer and the Internet will be excluded from participating. Also excluded will be individuals with life threatening medical illness, communicative disorder, lack of fluency in English, illiteracy, and major psychiatric conditions including psychoses, bipolar disorder, and alcohol or drug abuse. Patients will be required to add no medications to their regimen during the study period (approximately 6 weeks).

BASELINE ASSESSMENT. After reading and signing the informed consent, all participants will complete a baseline assessment consisting of questionnaires and a measure delivered by structured interview. Questionnaires will include the Health Assessment Questionnaire (HAQ), Quick Inventory of Depressive Symptomatology (QIDS), the PRIME-MD Somatic Symptoms Scale only (SSS), Positive and Negative Affect Scale (PANAS), Satisfaction with Life Scale (SWLS), and a demographics questionnaire. The structured interview will consist of the Composite International Diagnostic Interview (CIDI).

PROCEDURES: Subjects will be randomized to one of two groups. The psychological resilience building group's exercises will be posted on a state-of-the-art website known as "Authentic Happiness". Participants will be provided with the web address and shown how to access the site and the Research Portal where the 6 exercises that are the focus in this and other ongoing studies can be found. The journaling group will be instructed to write weekly for 60-minutes about how they used or plan to use their time over slightly varying time frames: 1) over the previous 24 hours, 2) over the previous week, 3) over the previous year, 4) in the next 24 hours, 5) in the next week and 6) in the next year. The journaling participants will use "PowerJournal". PowerJournal 0.2 for Windows is a downloadable program; once downloaded and installed on the computer, there is no further need for an Internet connection. This is a simple word-processing program, similar in style to Microsoft Word.

FOLLOW UP ASSESSMENT. After the intervention is complete, participants will be sent the same questionnaires (plus the Follow-Up Form) as used in the pre-intervention battery by mail and asked to return the questionnaires in the self-addressed, stamped envelope included. We estimate that these questionnaires will take about 30 minutes to complete. This will concluded their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Qualified patients will be primary care patients who meet the following inclusion and exclusion criteria: Patients between the ages of 18 and 75 seeking medical care for physical symptoms (i.e., persistent fatigue, pain complaints, and gastrointestinal, cardiovascular or musculoskeletal symptoms). No major medical illness to explain symptom(s) is found after detailed physical and laboratory assessment. Patients with common disorders such as hypertension, asthma, diabetes, low back strain, etc., will be included if in the opinion of the physician the presenting physical symptoms are not due to the underlying disorder. In order to enter the study, patients must meet criteria for at least 4 medically unexplained symptoms out of the 42 somatic symptoms listed in the Composite International Diagnostic Interview (CIDI) rated as currently present if males and at least 6 symptoms if females (Escobar's abridged criteria).

Exclusion Criteria:

* Patients without ready access to a computer and the Internet will be excluded from participating. Also excluded will be individuals with life threatening medical illness, communicative disorder, lack of fluency in English, illiteracy, and major psychiatric conditions including psychoses, bipolar disorder, and alcohol or drug abuse. Patients will be required to add no medications to their regimen during the study period (approximately 6 weeks).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptoms | Baseline and 6 weeks
Positive and Negative Affect Scale | Baseline and 6 weeks
Satisfaction with Life Scale | Baseline and 6 weeks

SECONDARY OUTCOMES:
Patient Health Questionnaire | Baseline and 6 weeks
Health Assessment Questionnaire | Baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Afton L Hassett, Psy.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ-Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

REFERENCES:
- See also: Robert Wood Johnson Medical School — http://rwjms.umdnj.edu/